CLINICAL TRIAL: NCT00655044
Title: Observational, Safety Study in Subjects Using Levemir® (Insulin Detemir) for the Treatment of Type 1 or Type 2 Diabetes Mellitus
Brief Title: Evaluation of Levemir® for the Treatment of Type 1 and 2 Diabetes
Acronym: PREDICTIVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3514
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 and type 2 diabetes patients
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Safety and effectiveness data collection in connection with the use of drug Levemir in daily clinical practice.
  Other Names: Levemir®; NN304

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to evaluate the incidence of serious adverse drug reactions while using Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes
* Candidates of use of a basal insulin as part of their diabetes regimen

Exclusion Criteria:

* Unwilling to adhere to therapy or follow up
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 and type 2 diabetes patients
Sampling Method: Non-Probability Sample
Enrollment: 3637 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
HbA1C | after 12 weeks

SECONDARY OUTCOMES:
Safety | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Moscow, Russia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com